CLINICAL TRIAL: NCT00682006
Title: Topical Application of Chlorhexidine to the Umbilical Cord for Prevention of Omphalitis and Neonatal Mortality in Rural District of Pakistan: A Community-based Randomized Control Trial
Brief Title: Topical Application of Chlorhexidine to the Umbilical Cord for Prevention of Omphalitis and Neonatal Mortality in Rural District of Pakistan
Acronym: Chlorhexidine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: John Snow, Inc. (Industry)
Responsible Party: Dr Zulfiqar A Bhutta, The Aga Khan University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 683-Ped/ERC-06
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Omphalitis
Keywords: Omphalitis; 4% Chlorhexidine; Newborns
MeSH Terms: interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): In this arm we recruited 2,400 subjects who received Intervention.
  Interventions: Drug: 4% Chlorhexidine
- B (Experimental): In this Arm, we recruited 2,400 subjects who received intervention.
  Interventions: Other: Hand washing Soap
- C (Experimental): In this Arm, we recruited 2,400 subjects who received intervention.
  Interventions: Drug: 4% Chlorhexidine
- D (No Intervention): In this Arm, we recruited 2,400 subjects for Observation and comparison. This was the prime control group.

INTERVENTIONS:
Drug: 4% Chlorhexidine — 4% Chlorhexidine was provided to be applied in this arm to Mothers through TBAs.
  Arms: A
Other: Hand washing Soap — Hand washing soap was provided to Mothers through TBAs.
  Arms: B
Drug: 4% Chlorhexidine — 4% Chlorhexidine was provided to be applied by Mothers through TBAs.
  Arms: C

SUMMARY:
The investigators hypothesize that application of 4% Chlorhexidine to the cord stump and meticulous hand washing by primary health care providers of newborn infants will reduce the incidence of Omphalitis and thereby Neonatal Mortality as compared to standardized dry cord care.

DETAILED DESCRIPTION:
The prime objective of this study is to estimate the independent effect of 4% Chlorhexidine solution application to cord stump and hand washing with soap by mothers of newborns for 2 weeks after birth in reducing Omphalitis in neonates compared to routine cord care by TBAs (Traditional Birth Attendant) in rural district of Sindh, Pakistan.

This study will be conducted in existing health infrastructure in a community setting with the help of two principal health care providers, TBAs and CHWs Community Health Workers) involved in maternal and newborn care. The TBAs conducting delivery wil be trained to wash hands with soap and water after completion of delivery and apply chlorhexidine to the Umbilical Cord Stump. The procedure will be repeated by the mother on the subsequent days up til 14 days from birth. The CHWs will also be trained to recognized signs of Omphalitis and record Cord Care in a systemic manner in a structured proforma.

The study will continue longitudinally for a period of one year to follow newborn for the signs of Omphalitis.

ELIGIBILITY:
Inclusion Criteria:

* All healthy newborns, born in the study setting will be systematically enrolled in the trial

Exclusion Criteria:

* Infants with congenital/birth defects
* Infants with any localized infection on the peri-umbilical region at the time of birth or application of any other material such as dung, etc before enrollment on the Cord.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9800 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Neonatal Omphalitis | By the end of the styudy
Rate of Neonatal Mortality | By the end of the Study

SECONDARY OUTCOMES:
Breastfeeding rate | By the end of the Study
Rate of Serious Neonatal Infections | By the end of the Study
Utilization of Clean Delivery Kits | By the end of the Study
Application Practice of Chlorhexidine | By the end of the Study

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar Dr Bhutta, MBBS, PhD, FRCP, MRCP, Principal Investigator — Aga Khan University
Locations (1):
- Proejct Office, Dadu, Sindh, Pakistan

REFERENCES:
- [Derived] Soofi S, Cousens S, Imdad A, Bhutto N, Ali N, Bhutta ZA. Topical application of chlorhexidine to neonatal umbilical cords for prevention of omphalitis and neonatal mortality in a rural district of Pakistan: a community-based, cluster-randomised trial. Lancet. 2012 Mar 17;379(9820):1029-36. doi: 10.1016/S0140-6736(11)61877-1. Epub 2012 Feb 8. PMID 22322126